CLINICAL TRIAL: NCT06129903
Title: The Effect of Enhanced Behavioral Healthcare on Self-Reported Depression, Anxiety, and Health-Related Quality of Life Among Patients With Musculoskeletal Sarcoma Undergoing Surgery: A Randomized Pilot Study
Brief Title: Study Assessing the Effects of Early Psychiatric Referral on Mental Health and Quality of Life in People With Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-247
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Sarcoma; Bone Sarcoma; Soft Tissue Sarcoma
Keywords: Sarcoma; Bone Sarcoma; Soft Tissue Sarcoma; Quality of Life; 23-247; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Masks; Behavioral Sciences

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Psychiatric Referral (Experimental): Participants will be randomized to the Early Psychiatric Referral group
  Interventions: Other: referral to the Memorial Sloan-Kettering Cancer Center (MSK) Department of Psychiatry and Behavioral Sciences.
- No Referral (No Intervention): Participants will be randomized to the No Referral group

INTERVENTIONS:
Other: referral to the Memorial Sloan-Kettering Cancer Center (MSK) Department of Psychiatry and Behavioral Sciences. — The primary intervention in this study is referral to the Memorial Sloan-Kettering Cancer Center (MSK) Department of Psychiatry and Behavioral Sciences. This study will not dictate specific psychiatry interventions beyond providing the referral.
  Arms: Early Psychiatric Referral

SUMMARY:
The purpose of this study is to investigate the feasibility of early access to mental healthcare during sarcoma treatment as well as to assess the association between early access to psychiatric care and depression, anxiety, postoperative outcomes, and patient satisfaction in patients undergoing surgery for musculoskeletal sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Tissue diagnosis of primary bone or soft tissue sarcoma

  o Note: high suspicion of sarcoma on history and imaging acceptable, if reviewed and approved by the PI
* Presenting to the Orthopaedic Surgery Service
* Treatment plan includes surgery at MSK for treatment of the primary sarcoma
* No previous treatment for sarcoma
* Proficient in English

  * As determined by use of the Census-LEP question
  * The patient's response to the question: "How well do you speak English?" must be "very-well" for inclusion. Additionally, English must be identified as the patient's preferred language for discussing healthcare.

Exclusion Criteria:

* Significant psychiatric disturbance determined from self-report and/or chart review, sufficient, in the investigator's judgment, to preclude participation in the study" (e.g., underlying severe mental illness, h/o suicide attempts, or h/o psychiatric admissions) Clinical concern at the time of randomization of mental health urgency or emergency requiring evaluation; urgency and emergency will be defined as moderate or high scores, respectively, on the CSSR-S or according to the judgment of the orthopaedic physician evaluating the patient
* Note: investigators considered exclusion of patients with no or mild symptoms of anxiety and depression, however due to risk of new symptoms arising during the course of treatment, risk of underreporting, risk of under detection, and given prior data on the high prevalence of symptoms, we elected to include all patients in this pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-11-07 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
The number of participants who complete scheduled study visits | 2 years
  The study will evaluate the feasibility of conducting a randomized clinical trial studying the impact of early referral to psychiatry (versus no referral) on depression and anxiety symptoms in patients with musculoskeletal sarcoma by examining the rates of eligibility, acceptance, uptake rate, and adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Bartelstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York
  - William Beaumont Army Medical Center, Fort Bliss, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org